CLINICAL TRIAL: NCT01313273
Title: Randomised, Phase III Multicenter, Open Study of Lanreotide in Non Metastatic Castration-resistant Prostate Cancer Patients Presenting Elevated Chromogranin A Levels
Brief Title: Study of Lanreotide in Non Metastatic Castration-resistant Prostate Cancer Patients
Acronym: POSEIDON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrolment
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-93-52030-738; 2010-019862-10 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other)
  Interventions: Drug: Non steroidal anti androgens and LHRH-a
- Arm B (Experimental)
  Interventions: Drug: Lanreotide, non steroidal anti androgens and LHRH-a

INTERVENTIONS:
Drug: Lanreotide, non steroidal anti androgens and LHRH-a — Lanreotide 120 mg. Injection every 28 days, to be administered till progression or for a maximum of 24 months.
  Non steroidal anti androgens (e.g. bicalutamide 50 mg/day to be administered till progression) plus LHRH-a (e.g. triptorelin 3.75 mg/month till progression.
  Arms: Arm B
Drug: Non steroidal anti androgens and LHRH-a — Non steroidal anti androgens (e.g. bicalutamide 50 mg/day to be administered till progression) plus LHRH-a (e.g. triptorelin 3.75 mg/month till progression
  Arms: Arm A

SUMMARY:
The aim of the study is to compare in an exploratory fashion the efficacy on progression-free survival of lanreotide in addition to non steroidal anti androgens and LHRH-a in non metastatic castrate resistant prostate cancer patients.

DETAILED DESCRIPTION:
LHRH-a=Luteinizing Hormone-Releasing Hormone Analogues

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of prostate cancer
* Evidence of PSA progression despite castrate levels of testosterone (<50 ng/dL) following orchiectomy or during therapy with luteinizing hormone releasing hormone agonists (LHRH-a)
* Patients with non-metastatic or stable metastatic disease
* Chromogranin A elevation above normal range (confirmed by a second evaluation at least 1 week later) [cut off levels will be > 20 U/L for enzyme linked immunosorbent (ELISA) assay and > 100 ng/ml for immunoradiometric (IRMA) assay]

Exclusion Criteria:

* Patients who according to the investigator opinion are candidates to be treated immediately with chemotherapy (e.g. docetaxel)
* First line treatment with antiandrogen in monotherapy
* Visceral metastasis
* Previous or concomitant treatment with a somatostatin analogue

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- A.O. S. Luigi Gonzaga, Orbassano ( TO), Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects ≥18 years meeting inclusion criteria were recruited for this study.
Pre-assignment Details: Investigators screened 8 subjects. Randomised 3 subjects and 5 were not randomised.
Groups:
- Arm A: Non-steroidal Anti Androgens + LHRH-a: Non-steroidal anti androgens (e.g. bicalutamide 50 mg/day) plus Luteinizing Hormone-Releasing Hormone Analogues (LHRH-a) (e.g. triptorelin 3.75 mg/month) till progression.
- Arm B: Lanreotide + Non Steroidal Anti Androgens and LHRH-a: Lanreotide 120 mg injection every 28 days till progression or for a maximum of 24 months plus non steroidal anti androgens (e.g. bicalutamide 50 mg/day) and LHRH-a (e.g. triptorelin 3.75 mg/month) till progression.
Period: Overall Study
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non Steroidal Anti Androgens and LHRH-a
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — INCLUSION CRITERIA 4 NOT RESPECTED | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Screening Chromogranin A-in normal range | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Non-steroidal Anti Androgens + LHRH-a: Non-steroidal antiandrogens (e.g. bicalutamide 50 mg/day) plus LHRH-a (e.g. triptorelin 3.75 mg/month) till progression.
- Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a: Lanreotide 120 mg injection every 28 days till progression or for a maximum of 24 months plus non-steroidal antiandrogens (e.g. bicalutamide 50 mg/day) and LHRH-a (e.g. triptorelin 3.75 mg/month) till progression.
- Total: Total of all reporting groups
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 72.50 [61.00 to 84.00] | 57.00 [57.00 to 57.00] | 61.00 [57.00 to 84.00]
Age, Customized [Number; unit: Participants]
  >=65 years | 1 | 0 | 1
  Between 18 and 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Italy | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: Week 96
Population: Study early terminated due to poor enrollment.
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Prostate Specific Antigen (PSA) Response
Time Frame: Week 96
Population: Study early terminated due to poor enrollment
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Median Time to PSA Response
Time Frame: Week 96
Population: Study early terminated due to poor enrollment
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Reduction in Chromogranin A Serum Levels
Time Frame: Baseline, Week 96
Population: Study early terminated due to poor enrollment
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were reported from Baseline (visit 2) to visit 10 (week 96 - End of study)
Description: All Adverse Events (AEs) documented for this study were treatment emergent. Overall, for 1 patient (100.0%) of Arm B at least one AE, at least one AE related to study treatment and at least one severe AE were reported.
Arm/Group | Arm A: Non-steroidal Anti Androgens + LHRH-a | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Non-steroidal Anti Androgens + LHRH-a (N=2) | Arm B: Lanreotide + Non-steroidal Antiandrogens and LHRH-a (N=1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3)
Transaminases increased (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No